CLINICAL TRIAL: NCT07159698
Title: Clinical Profile of a Patient After Myocardial Infarction and Acute Cerebrovascular Accident Based on Outpatient Register Data
Brief Title: Clinical Profile of a Patient After MI and ACVA Based on Outpatient Register Data
Status: Enrolling by invitation | Type: Observational
Sponsor: State Institution "Republican Scientific and Practical Center" Cardiology, Belarus (Other)
Collaborators: Belarusian State Medical University (Other)
Responsible Party: Principal Investigator, Pabivantsava Natallia, Head of the Laboratories of Comorbid Cardiology, RSPC Cardiology, Ph.D (Medicine), State Institution "Republican Scientific and Practical Center" Cardiology, Belarus
Other Study IDs: 20250326
Record Dates: First submitted 2025-08-06; First posted 2025-09-08 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Acute Cerebrovascular Accident; Myocardial Infarction (MI)
Keywords: register; myocardial infarction; acute cerebrovascular accident; quality of medical care; outpatient and polyclinic institutions
MeSH Terms: conditions — Stroke; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- myocardial infarction (MI): Patients with a history of MI of any remoteness; visit to the outpatient clinic for any reason during the period from January 1, 2019, to December 31, 2022; age 18 years or older; the presence of informed consent for the processing of personal data in the outpatient medical record; and permanent residence in the city where the register is being established.
- acute cerebrovascular accident (ACVA): Patients with a history of ACVA of any remoteness; visit to the outpatient clinic for any reason during the period from January 1, 2019, to December 31, 2022; age 18 years or older; the presence of informed consent for the processing of personal data in the outpatient medical record; and permanent residence in the city where the register is being established.
- acute cerebrovascular accident + myocardial infarction (ACVA+MI): Patients with a history of MI and ACVA of any remoteness; visit to the outpatient clinic for any reason during the period from January 1, 2019, to December 31, 2022; age 18 years or older; the presence of informed consent for the processing of personal data in the outpatient medical record; and permanent residence in the city where the register is being established.

SUMMARY:
This is a retrospective observational study using the methodology of creating medical registries. The expected number of patients included in the registry is about 2000 patients with myocardial infarction and/or ACVD of any duration and concomitant non-cardiac diseases of therapeutic profile in pilot healthcare organizations for any reason during 2019-2022 based on the source medical records data.

DETAILED DESCRIPTION:
Abstract The article presents the results of the analysis of outpatient register data of patients after myocardial infarction (MI) and acute cerebrovascular accident (ACVA). Based on the epidemiological characteristics of individuals included in the register, a clinical "portrait of a patient" after an acute cardiovascular event was formed. The features of clinical and laboratory parameters, as well as behavioral and metabolic factors of cardiovascular risk in patients included in the study were determined; and adherence to treatment before and after the reference event was assessed over a 12-year follow-up period.

The objective of the study: to determine the features of clinical and epidemiological characteristics and parameters of laboratory and instrumental studies, the profile of cardiovascular risk factors in patients with a history of MI and ACVA, and to establish their adherence to treatment before and after the reference event over a 12-year follow-up period.

Materials and methods. The investigators analyzed the data of 410 patients who applied to an outpatient and polyclinic healthcare organization between January 1, 2019, and December 31, 2022, with confirmed acute (recurrent) myocardial infarction and/or cerebral infarction that occurred between January 1, 2010, and December 31, 2019. Patients were included in the register after establishing their vital status as of January 1, 2020. The data of records and reports from healthcare organizations (forms 025/u, 131-u) and electronic outpatient records of medical information systems (MIS) from outpatient polyclinic institutions (OPI) were used. The results of the retrospective stage analysis of the study and the electronic patient database from the information and analytical system "Register of MI/ACVA" were presented. Standard methods of descriptive and analytical statistics, statistical software packages (SPSS, SAS, STATISTIKA 10, Stata) and programming languages (R, Python) were used.

ELIGIBILITY:
Inclusion Criteria:

* history of MI and/or ACVA of any remoteness;
* visit to the outpatient clinic for any reason during the period from January 1, 2019, to December 31, 2022;
* age 18 years or older;
* the presence of informed consent for the processing of personal data in the outpatient medical record;
* permanent residence in the city where the register is being established.

Exclusion Criteria:

* non-compliance with the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who applied to the outpatient clinic for any reason between 2019-2022 in order to identify and "look for" patients after acute cardiovascular event and myocardial infarction, meeting the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1520 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Identification of the main risk factors for the development of heart attacks and/or strokes in the group of studied patients. | 5 years
  For this purpose, primary medical documentation and patient's dispensary observation cards were used. Participants achieved target levels of indicators of the main risk factors according to established standards in accordance with international recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Grigorenko, Ph.D, Study Chair — Republican Scientific and Practical Center of Cardiology
Locations (1):
- Republican Scientific and Practical Center of Cardiology, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: Undecided
Protection of personal data

DOCUMENTS (1):
  • Study Protocol (2025-09-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT07159698/Prot_000.pdf